CLINICAL TRIAL: NCT02957084
Title: Anatomic Features of the Neck and Preoperative Tests as Predictive Markers of Difficult Direct Laryngoscopy
Brief Title: Anatomic Features of the Neck and Preoperative Tests as Predictive Markers of Difficult Laryngoscopy
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Chara Liaskou, RN, Msc, Phd(c), National and Kapodistrian University of Athens
Other Study IDs: 10634
Record Dates: First submitted 2016-10-29; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Airway Management; Predictive Value of Tests
Keywords: difficult laryngoscopy; neck circumference; sternomental distance; thyromental distance; hyomental distance; thyrosternal distance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this prospective, open cohort study the diagnostic value of tests based on neck anatomy in predicting difficult laryngoscopy was assessed.

The anatomic features of the neck measured were head extension, mouth opening, upper lip bite, Mallampati class, thyromental distance, sternomental distance, ratio of height to thyromental, neck circumference, thyrosternal distance, hyomental distance at full head extension (FHE) and at neutral position (NP), ratio of neck circumference to thyromental distance and ratio of hyomental distance FHE to hyomental distance NP.

DETAILED DESCRIPTION:
Difficult airway assessment is based on various anatomic parameters of upper airway, much of it being concentrated on oral cavity and the pharyngeal structures. The diagnostic value of tests based on neck anatomy in predicting difficult laryngoscopy was assessed in this study .

The sample consisted of adult patients scheduled to receive general anaesthesia. Anatomic features of the neck were measured pre-operatively.

The anatomic features of the neck measured were thyromental distance, sternomental distance, ratio of height to thyromental, neck circumference, thyrosternal distance, hyomental distance at full head extension (FHE) and at neutral position (NP), ratio of neck circumference to thyromental distance and ratio of hyomental distance FHE to hyomental distance NP. The commonly used predictive tests head extension, mouth opening, upper lip bite test and Mallampati class were also measured.

The laryngoscopic view was classified according to the Cormack-Lehane Grade (1-4). Difficult laryngoscopy was defined as Cormack-Lehane Grade 3 or 4. Years of experience of the anaesthesiologists were recorded, as well as the number of tries needed to intubate the patient.

The optimal cut-off points for each predictive tests were identified by using receiver operating characteristic analysis. Sensitivity, specificity and positive predictive value and negative predictive value (NPV) were calculated for each test. Multivariate analysis with logistic regression, including all variables, was used to create a predictive model. Comparisons between genders were also performed to explore possible differences in diagnostic value and cut-off points. Finally, the years of experience of the clinician and the number of tries needed to intubate the patient were compared to assess risk of bias.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* BMI less than 35 kg/m2
* No known neck or airway pathology
* Scheduled for surgical procedures under general anaesthesia with tracheal intubation

Exclusion Criteria:

* Age less than 18 years
* BMI higher than 35 kg/m2
* Obvious airway malformations
* Need for rapid sequence induction/intubation under cricoid pressure
* Awake intubation
* Cervical spine pathology requiring specific manipulation
* Obstetric cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with BMI less than 35 kg/m2, wihthout any known neck or airway pathology, scheduled for surgical procedures under general anaesthesia with tracheal intubation were assessed for eligibility to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1142 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difficult laryngoscopy classification using Cormack-Lehane Grade | immediate
  Assessment of difficult laryngoscopy at the time of the airway management procedure. Classified as Grade I - visualization of entire laryngeal aperture, grade II - visualization of only posterior commissure of laryngeal aperture, grade III - visualization of only epiglottis, grade IV - visualization of just the soft palate.

SECONDARY OUTCOMES:
Thyromental distance measured in cm with a measuring tape | immediate
  The distance from the mentum to the thyroid notch while the patient's neck is fully extended and the mouth closed
Sternomental distance measured in cm with a measuring tape | immediate
  The distance from the suprasternal notch to the mentum while the patient's neck is fully extended and the mouth closed
Ratio of height to thyromental distance | immediate
  Calculated ratio of the height in cm to the aforementioned thyromental distance
Thyrosternal distance calculated in cm | immediate
  Calculated from the subtraction: sternomental (cm) minus thyromental (cm)
Neck circumference measured in cm with a measuring tape | immediate
  Measurement at the level of the cricoid cartilage while the patient's neck is in neutral position
Ratio of neck circumference to thyromental distance | immediate
  Calculated ratio of the neck circumference to the aforementioned thyromental distance
Hyomental distance at full head extension (FHE) measured in cm with a measuring tape | immediate
  The distance from the mentum to the hyoid bone while the patient's neck is fully extended and the mouth closed
Hyomental distance at neutral position (NP) measured in cm with a measuring tape | immediate
  The distance from the mentum to the hyoid bone while the patient's neck is in neutral position and the mouth closed
Ratio of hyomental distance at FHE to hyomental distance at NP | immediate
  Calculated ratio of the aforementioned variables
Mallampati class | immediate
  Classified as class I - soft palate, fauces, uvula, and pillars seen, class II - soft palate, fauces, and uvula seen, class III - soft palate and base of uvula seen and class IV - soft palate not visible.
Mouth opening measured in cm with a measuring tape | immediate
  The distance between the upper and lower incisors with the mouth fully open
Upper lip bite test | immediate
  Classified as class I - lower incisors can bite the upper lip above the vermilion line, class II - lower incisors can bite the upper lip below the vermilion line and class III - lower incisors cannot bite the upper lip.
Head extension measured in degrees with goniometer | immediate
  The patient was asked to hold head erect, facing directly to the front, then asked to extend the head maximally and the examiner estimated the angle traversed by the occlusal surface of upper teeth using a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Chryssoula Staikou, MD, PhD, Assistant Professor, Study Director — National and Kapodistrian University of Athens, 1st Department of Anaesthesia, Aretaieio Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frova G, Sorbello M. Algorithms for difficult airway management: a review. Minerva Anestesiol. 2009 Apr;75(4):201-9. Epub 2008 Oct 23. PMID 18946426
- [Background] Cheney FW. The American Society of Anesthesiologists Closed Claims Project: what have we learned, how has it affected practice, and how will it affect practice in the future? Anesthesiology. 1999 Aug;91(2):552-6. doi: 10.1097/00000542-199908000-00030. No abstract available. PMID 10443619
- [Background] Chipas A, Ellis W, Zaglaniczny K. Airway management. In: Zaglaniczny K, Nagelhout J. Nurse Anesthesia. 3rd edition. USA: Elsevier Saunders; 2004:408
- [Background] Crosby ET, Cooper RM, Douglas MJ, Doyle DJ, Hung OR, Labrecque P, Muir H, Murphy MF, Preston RP, Rose DK, Roy L. The unanticipated difficult airway with recommendations for management. Can J Anaesth. 1998 Aug;45(8):757-76. doi: 10.1007/BF03012147. PMID 9793666
- [Background] Lundstrom LH. Detection of risk factors for difficult tracheal intubation. Dan Med J. 2012 Apr;59(4):B4431. PMID 22459727
- [Background] Peterson GN, Domino KB, Caplan RA, Posner KL, Lee LA, Cheney FW. Management of the difficult airway: a closed claims analysis. Anesthesiology. 2005 Jul;103(1):33-9. doi: 10.1097/00000542-200507000-00009. PMID 15983454
- [Background] Rucker JC, Cole D, Guerina LR, Zoran N, Chung F, Friedman Z. A prospective observational evaluation of an anatomically guided, logically formulated airway measure to predict difficult laryngoscopy. Eur J Anaesthesiol. 2012 May;29(5):213-7. doi: 10.1097/EJA.0b013e3283502168. PMID 22450528
- [Background] Shiga T, Wajima Z, Inoue T, Sakamoto A. Predicting difficult intubation in apparently normal patients: a meta-analysis of bedside screening test performance. Anesthesiology. 2005 Aug;103(2):429-37. doi: 10.1097/00000542-200508000-00027. PMID 16052126
- [Background] Koay CK. Difficult tracheal intubation--analysis and management in 37 cases. Singapore Med J. 1998 Mar;39(3):112-4. PMID 9632969
- [Background] Burkle CM, Walsh MT, Harrison BA, Curry TB, Rose SH. Airway management after failure to intubate by direct laryngoscopy: outcomes in a large teaching hospital. Can J Anaesth. 2005 Jun-Jul;52(6):634-40. doi: 10.1007/BF03015776. PMID 15983152
- [Background] Cattano D, Panicucci E, Paolicchi A, Forfori F, Giunta F, Hagberg C. Risk factors assessment of the difficult airway: an italian survey of 1956 patients. Anesth Analg. 2004 Dec;99(6):1774-1779. doi: 10.1213/01.ANE.0000136772.38754.01. PMID 15562070
- [Background] Rose DK, Cohen MM. The airway: problems and predictions in 18,500 patients. Can J Anaesth. 1994 May;41(5 Pt 1):372-83. doi: 10.1007/BF03009858. PMID 8055603
- [Background] Turkan S, Ates Y, Cuhruk H, Tekdemir I. Should we reevaluate the variables for predicting the difficult airway in anesthesiology? Anesth Analg. 2002 May;94(5):1340-4, table of contents. doi: 10.1097/00000539-200205000-00055. PMID 11973217
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Background] Khan ZH, Kashfi A, Ebrahimkhani E. A comparison of the upper lip bite test (a simple new technique) with modified Mallampati classification in predicting difficulty in endotracheal intubation: a prospective blinded study. Anesth Analg. 2003 Feb;96(2):595-9, table of contents. doi: 10.1097/00000539-200302000-00053. PMID 12538218
- [Background] Patil VU, Stehling LC, Zauder HL. Predicting the difficulty of intubation utilizing an intubation gauge. Anesthesiol Rev. 1983;10:32-3.
- [Background] Savva D. Prediction of difficult tracheal intubation. Br J Anaesth. 1994 Aug;73(2):149-53. doi: 10.1093/bja/73.2.149. PMID 7917726
- [Background] Naguib M, Malabarey T, AlSatli RA, Al Damegh S, Samarkandi AH. Predictive models for difficult laryngoscopy and intubation. A clinical, radiologic and three-dimensional computer imaging study. Can J Anaesth. 1999 Aug;46(8):748-59. doi: 10.1007/BF03013910. PMID 10451134
- [Background] Gupta S, Sharma R, Jain D. Airway assessment: predictors of difficult airway. Indian J Anaesth. 2005:49(4):257-62
- [Background] Schmitt HJ, Kirmse M, Radespiel-Troger M. Ratio of patient's height to thyromental distance improves prediction of difficult laryngoscopy. Anaesth Intensive Care. 2002 Dec;30(6):763-5. doi: 10.1177/0310057X0203000607. PMID 12500514
- [Background] Huh J, Shin HY, Kim SH, Yoon TK, Kim DK. Diagnostic predictor of difficult laryngoscopy: the hyomental distance ratio. Anesth Analg. 2009 Feb;108(2):544-8. doi: 10.1213/ane.0b013e31818fc347. PMID 19151285
- [Background] Greek Society for Airway management, Basic and Advanced Management of the Airway, 2nd edition, Athens, 2011